CLINICAL TRIAL: NCT04269564
Title: the Use of Intraoperative Bedside Lung Ultrasound in Optimizing "Positive End Expiratory Pressure"PEEP in Patients Undergoing Laparoscopic Bariatric Surgeries
Brief Title: Optimizing PEEP in Laparoscopic Bariatric Surgery Using Bedside Lung Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohamed abdel ghany ali, Anesthesia lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MS-263-2019
Record Dates: First submitted 2020-02-03; First posted 2020-02-17 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Atelectasis, Postoperative Pulmonary
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (No Intervention): Group A patients received the standard ventilation protocol as follows: volume-controlled ventilation mode, with VT 6 ml/kg of ideal body weight, inspiratory : expiratory ratio 1 : 2, a PEEP of 4 cmH2O, and respiratory rate 10-12 breaths/min that will be adjusted to keep end-tidal carbon dioxide tension (EtCO2) between 35 and 40 mmHg and inspired oxygen fraction of 0.5.
- group B (Active Comparator): Patients in group B received the standard ventilation protocol with stepwise peep until end of surgery and extubation.
  Interventions: Device: stepwise PEEP

INTERVENTIONS:
Device: stepwise PEEP — * a PEEP of 4 cmH2O will be used after intubation till 5 minutes after pneumoperitonium, and adjusted in a step wise approach after lung ultrasound by adding 2 cmH2O, repeating ultrasound 5 minutes after every change in peep till no lung collapse is detected by lung ultrasound with a maximal peep of 10 cmH2O, or if hemodynamic instability occurs.
  * Lung ultrasound examination will be performed at a minimum three times in each patient; the first will be performed 1 min after starting mechanical ventilation of the lungs, 5 minutes after pneumoperitonium, 5 min after every peep increase in stepwise peep group and the last time at the end of the surgery.
  We define anaesthesia-induced atelectasis to be significant if any region has a consolidation score of ≥ 2.
  Arms: group B

SUMMARY:
Lung ultrasound imaging is a promising non-invasive, non-radiant, portable and easy to use tool that as yet to be studied in the intraoperative setting.

in our current study, we are trying to reach the optimum PEEP in laparoscopic bariatric patients to prevent postoperative collapse and atlectasis with simple non-invasive procedure.

ELIGIBILITY:
Inclusion Criteria:

* they are between 18 and 65 years of age
* BMI more than 35
* patients with normal respiratory functions
* ASA 1 or 2

Exclusion Criteria:

* Previous lung surgery
* Bronchial asthma
* Contralateral lung bullae 4. Uncompensated cardiac disease (NYHA class 3 or 4) 5. Obstructive or restrictive lung disease 6. Patients on home oxygen therapy 7. Hemodynamic instability and increased intracranial pressure 8. In adittion , any patient who developes hemodynamic instability (MAP <60mmHg) or hypoxia (Po2 less than 60) during the study will excluded from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2020-08-19 (Actual)

PRIMARY OUTCOMES:
efficacy of lung ultrasound in optimizing peep | intraoperative and early postoperative first 24 hours after recovery from anaesthesia
  to evaluate the effect of lung ultrasound in optimizing peep in obese patients undergoing laparoscopic surgeries on the Incidence of intraoperative hypoxia and atlectasis

SECONDARY OUTCOMES:
effect on early postoperative oxygenation | 24 hours postoperative
  Evaluating the effect of stepwise PEEP approach on the incidence of early postoperative in the first 24 hours atelectasis and oxygenation.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Cairo, Egypt

REFERENCES:
- [Background] Chooi YC, Ding C, Magkos F. The epidemiology of obesity. Metabolism. 2019 Mar;92:6-10. doi: 10.1016/j.metabol.2018.09.005. Epub 2018 Sep 22. PMID 30253139
- [Background] Lobo B, Hermosa C, Abella A, Gordo F. Electrical impedance tomography. Ann Transl Med. 2018 Jan;6(2):26. doi: 10.21037/atm.2017.12.06. PMID 29430443
- [Background] Monastesse A, Girard F, Massicotte N, Chartrand-Lefebvre C, Girard M. Lung Ultrasonography for the Assessment of Perioperative Atelectasis: A Pilot Feasibility Study. Anesth Analg. 2017 Feb;124(2):494-504. doi: 10.1213/ANE.0000000000001603. PMID 27669555